CLINICAL TRIAL: NCT04131400
Title: Establishment of the National Registry for Inherited Retinal Dystrophy in Iran
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Head of department, Shahid Beheshti University of Medical Sciences
Other Study IDs: 2222
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Inherited Retinal Dystrophy Primarily Involving Sensory Retina; Inherited Retinal Dystrophy Primarily Involving Retinal Pigment Epithelium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Inherited Retinal Dystrophy: known patients with a diagnosis of inherited retinal dystrophy (IRD) will be recruited to identify the type of IRD diagnosis. The comprehensive ophthalmic examinations and retinal imaging will be performed. Additionally, blood sample of all participants and their family members will be kept in our bio- bank for genetic testing.
  Interventions: Diagnostic Test: Visual Acuity Testing and Retinal Imaging

INTERVENTIONS:
Diagnostic Test: Visual Acuity Testing and Retinal Imaging — All clinical and para- clinical tests including visual acuity assessment, perimetry, optical coherence tomography (OCT), enhanced depth- OCT, OCT angiography, color fundus, autofluorescence and infrared fundus photography will be performed

SUMMARY:
Purpose: To establish of the national Inherited Retinal Dystrophy Registry (IRDR) in Iran.

Methods: This study is a community-based participatory research that is approved by the Ministry of Health and Medical Education of Iran in 2016. To provide the minimum data set (MDS), several focus group meetings will be held with participation of the faculty members of the Ophthalmic Research Center affiliated to Shahid Beheshti University of Medical Sciences (SBMU). Final MDS will be presented to the software engineering team to develop a web-based software. In the pilot phase, software will be set up in two referral centers including Labbafinejad Medical Center (Tehran) and Alzahra Eye Hospital (Zahedan) to discover the possible drawbacks. Final diagnosis will be made based on both clinical manifestations as well as genetic findings.The steering committee meetings are planned to be held each year with the presence of delegates of all centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a definite diagnosis of IRD diagnoses based on clinical examinations and genetic testing.

Exclusion Criteria:

* Individuals who have a suspected diagnosis of IRD disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: An initial registration will be performed only for subjects who has a diagnosis of IRD based on clinical and retinal imaging by an expert retina specialist, but definite diagnosis will be confirmed by genetic testing.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
prevalence and incidence of the different types of inherited retinal dystrophy in different regions of Iran. | 4 years
  The present study is designed to determine the prevalence and incidence of IRD diagnoses in different regions of Iran based on the crude data which will be registered in the Iranian IRD registry.

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran